CLINICAL TRIAL: NCT06112184
Title: A Prospective, Single-arm, Feasibility Study to Evaluate the Performance of the SK-M11/3A1 Digital Health Program With Participants Using an Autoinjector
Brief Title: Digital Health Program With Participants Using an Autoinjector
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidekick Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SK-M11/3A1-001
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Immune-Mediated Inflammatory Disease
Keywords: self-injection; digital solution; lifestyle change; disease education; medication adherence; immune-mediated inflammatory disease; IMID; healthy lifestyle
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: A prospective, single-arm, feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): All participants will use the SK-M11/3A1 digital health program for 12 weeks.
  Interventions: Other: SK-M11/3A1 Digital health program

INTERVENTIONS:
Other: SK-M11/3A1 Digital health program — Digital Health program with participants using an autoinjector delivered via the Sidekick mobile application (app)
  Other Names: SK-M11/3A1 Master your treatment

SUMMARY:
This is a prospective, single-arm, feasibility study. Up to thirty (30) participants meeting study eligibility criteria will use the SK-M11/3A1 digital health program for 12 weeks. The program will be delivered via the Sidekick mobile application (app).

The study objective is to evaluate the performance and safety of the SK-M11/3A1 digital health program when added to routine medical treatment of patients with Immune-Mediated Inflammatory Disease (IMID). All participants are using a prescribed medication for regular subcutaneous injection provided in a prefilled autoinjector.

DETAILED DESCRIPTION:
Numerous therapies are formulated for subcutaneous injections, enabling patients and caregivers to administer them at home instead of intravenously in-clinic. Despite the notable benefit and decrease in the treatment burden, the act of self-injecting and at-home administration inevitably imposes a substantial responsibility and burden on the patient.

To support the efforts to improve medication adherence and make the process of self-injecting more user friendly and easy, Sidekick Health (SKH) has developed a digital health program designed specifically for this purpose (SK-M11). SKH has paired this with disease-specific content that is indicated for patients with an Immune-Mediated Inflammatory Disease (IMID) (SK-3A1), addressing some of the most common challenges these patients encounter, as well as general assistance with making healthy lifestyle choices.

The aim of this study is primarily to assess the acceptability and feasibility of combining the SK-M11 and SK-3A1 and adding the digital health program to the Standard of Care (SoC) by measuring participants engagement, retention and satisfaction. Up to 30 IMID patients using a prescribed medication for regular subcutaneous injection provided in a prefilled autoinjector for self-injection in the home environment will be included. The participants will use SK-M11/3A1 for the study period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Patients diagnosed with IMID and already using or initiating an IMID therapy with a medicine for regular subcutaneous injection provided in a prefilled autoinjector for self-injection in the home environment, as prescribed by their doctor.
* Owns a smartphone compatible with the SK-M11/3A1 digital health program and is willing and able to use it
* Participant has been informed of the nature of the study and has been provided with electronic informed consent approved by the appropriate Independent Ethics Committee (IEC)
* Willing and able to comply with all protocol-specified items (app use, all scheduled visits, and completing questionnaires/surveys)

Exclusion Criteria:

* The patient has other concurrent conditions that in the opinion of the Investigator may compromise patient safety or study objectives
* Pregnant and/or breastfeeding females (self-reported) at baseline or during the course of the study (12 weeks)
* Enrollment in a concurrent study in which the study treatment may confound the evaluation of the investigational program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Retention/Engagement - completion | 12 weeks
  Percentage of users that complete the program. Completion is defined as finishing 75% of the program (9/12 weeks).
Retention/Engagement - activity | 12 weeks
  Percentage of active users throughout the program. Active is defined as visiting the app at least once per week.
Usability of the app | 12 weeks
  Average score of the Mobile Health App Usability Questionnaire (MAUQ) at end of program.
  The MAUQ is a self-administered questionnaire that has three subscales and is composed of in total 21 questions with a Likert scale of 7 options where 1 represents "strongly agree" to 7 "strongly disagree". Scores on the MAUQ range from 21 to 147, with a higher score representing better usability.

SECONDARY OUTCOMES:
Assessment of self-injection experience | 12 weeks
  Changes in self-reported scores (from Baseline to Week 12) as measured by the Self-Injection Assessment Questionnaire (SIAQ).
  The SIAQ is a self-reported questionnaire that is divided into pre- and post-study modules and for the purpose of this study, only the pre-study module is used. It is composed of 7 questions with a Likert scale of 5 options. For questions 1 to 6 a score of 1 represents "not at all" to 5 "extremely". For question 7 a score of 1 represents "very dissatisfied" to 5 "very satisfied". Scores on the SIAQ range from 7 to 35, with a lower score representing a good self-injection experience.
Use of in-app reminders | 12 weeks
  Percentage of users actively using in-app reminders (% users reacting to reminders) and medication log (% users entering data relating to the medicine and dosing)
Compliance with medication regime | 12 weeks
  Changes in self-reported scores (from Baseline to Week 12) as measured by the 5-item Compliance Questionnaire for Rheumatology (CQR5).
  The CQR5 is composed of 5 questions with a Likert scale of 5 options where 1 represents "completely disagree" to 5 "completely agree". Scores on the CQR5 range from 5 to 25, with a lower score representing lower compliance.
Evaluate the impact of patient education | 12 weeks
  Change in self-reported score (from baseline to 12 weeks) as measured by the Health Education Impact Questionnaire (heiQ) score.
  The heiQ has 8 subscales and is composed of in total 42 questions with a Likert scale of 4 options where 1 represents "strongly disagree" to 4 "strongly agree". Scores on the heiQ range from 42 to 168, with a lower score representing a low impact on patient education.

CONTACTS AND LOCATIONS:
Overall Officials: Bárður L Sigurgeirsson, MD, PhD, Principal Investigator — Húðlæknastöðin
Locations (1):
- Húðlæknastöðin dermatology clinic, Kopavogur, Iceland

IPD SHARING:
Plan to Share IPD: No
Anonymized Individual Participant Data may be shared with other researchers for relevant research purposes following complementary ethical review and approval from the Ethical Review Board.